CLINICAL TRIAL: NCT06156800
Title: Is Radiation-before-pathology a Feasible Approach in the Palliative Oncology Setting? A Pragmatic Clinical Trial (RT-NOW)
Brief Title: Is Radiation-before-pathology a Feasible Approach in the Palliative Oncology Setting? A Pragmatic Clinical Trial
Acronym: RT-NOW
Status: Recruiting | Type: Observational
Sponsor: David Palma (Other)
Responsible Party: Sponsor-Investigator, David Palma, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: RT-NOW
Record Dates: First submitted 2023-11-07; First posted 2023-12-05 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Cancer
Keywords: Palliative Irradiation; Biopsy; Radiation Therapy; Pathology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
When a doctor suspects cancer, often a biopsy is taken for testing to confirm if cancer is present. Usually, doctors would wait for the results of a biopsy before delivering radiation, but this may lead to a patient having to wait for a treatment that he or she urgently needs.

With long wait times for biopsies in Canada, this may lead to symptoms and risks of complications from cancer in the meantime. Therefore, this study is being done to answer the following question: Is it safe and feasible to deliver radiation before obtaining a biopsy in a carefully selected group of patients who urgently need radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Willing to provide informed consent
* Palliative treatment intent: either metastatic or incurable locally advanced disease
* Tissue diagnosis is not required for determination of dose/fractionation scheme
* Recent cross-sectional imaging [for example - Computed Tomography (CT), Magnetic Resonance Imaging (MRI), Positron Emission Tomography/Computed Tomography (PET/CT)] of the area to be treated, done within the past 3 months
* Treating physician considers the pre-test probability of cancer greater than 95 percent based on clinical judgement and radiological findings.
* The patient has at least 1 site of cancer amenable to biopsy

  * As per standard practices, if the radiation oncologist will be radiating the only site available to biopsy, they should proceed with caution. Participants should only be enrolled on trial if the risk of harm from delaying Radiation Therapy (RT) significantly outweighs the risks of possible non-diagnostic tissue. If the participant may potentially be eligible for systemic therapy, the treating radiation oncologist should consult a medical oncologist for an opinion regarding the risks of non-diagnostic molecular testing. The weighing of these priorities should be thoroughly discussed with the participant and the discussion should be documented.
  * Reasons for radiating a participant with a single lesion prior to biopsy include:

    * Spinal cord compression (actual or impending) and inoperable
    * Brain metastasis with significant symptoms or neurologic deficits and inoperable
    * Other lesions causing neurologic deficit
    * Pulmonary lesion causing or threatening lung obstruction
    * Uncontrolled bleeding (including hemoptysis and hematuria)
    * Superior vena cava obstruction (actual or impending)
    * Limited upside to molecular testing, as determined by the medical oncologist (for example - participant unfit for available systemic therapies, limited options for systemic therapy)
* Radiation is considered urgent (for example - participant should receive radiation prior to biopsy date) o Urgent indications may include but are not limited to the reasons listed previously, as well as the following:

  * Painful metastases or primary lesion not adequately responding to analgesia
  * Symptomatic brain metastases
  * Bleeding
  * Impending pathologic fracture

Exclusion Criteria:

* Participant is potentially eligible for curative treatment
* Clinical suspicion of lymphoma o Some features may be suggestive of lymphoma, including fever or night sweats (for example - B symptoms excluding weight loss), or imaging showing well-defined, homogenous lymphadenopathy. These findings are not exclusion criteria specifically, but should be considered by the clinician in formulating their differential diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with convincing clinical/radiological evidence of cancer, ineligible for curative treatment and awaiting a biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Percent of Inappropriate Use of Radiation Therapy in Participants with Urgent Indications Treated Prior to Biopsy Results | 2 weeks after biopsy results
  The percentage of participants in whom management would have differed, based on the final pathology, if the pathology had been known prior to radiation therapy.
  Inappropriate use of radiation therapy is defined as:
  If a non-cancerous process was treated, Or, the use of radiation therapy was inappropriate in hindsight (for example, the participant would have clearly been better treated with alternative options).

SECONDARY OUTCOMES:
Histological Diagnostic Accuracy | 2 weeks after biopsy results
  Histological diagnostic accuracy is defined as the percentage of biopsies that yielded a histological diagnosis. This will include a comparison of diagnostic yield between biopsies done at radiated vs. non-radiated sites.
Molecular Testing Accuracy | 2 weeks after biopsy results
  Molecular testing accuracy is defined as the percentage of biopsies that yielded enough viable tissue for molecular testing/diagnosis.
Number of Biopsy Attempts Required | 2 weeks after biopsy
Biopsy Complication Rates | 2 weeks after biopsy
Time from Enrollment to First Fraction of Radiation Therapy | Within 1 year after enrollment
Time from Enrollment to Biopsy | Within 1 year after enrollment
Evidence of Radiation Effect in Biopsy | 2 weeks after biopsy results
Overall Survival | 1 year after enrollment
Edmonton Symptom Assessment System Revised Scores | 2 weeks after radiation therapy of 2 weeks after biopsy
  Participants will rate their symptoms on a scale of 1 to 10, 0 being the best and 10 being the worst.
  Examples of symptoms included in the Edmonton Symptom Assessment System revised are pain, tiredness, nausea, appetite, depression, and so on.

CONTACTS AND LOCATIONS:
Overall Officials: David Palma, MD, Principal Investigator — London Health Sciences Centre, Lawson Health Research Institute
Locations (1):
- London Regional Cancer Program, London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Young S, O'Neil M, Laba JM, Nguyen TK, Qu XM, Goodman CD, Bauman GS, Warner A, Cecchini M, Palma DA. Radiation-before-pathology approach in the palliative oncology setting: a pragmatic clinical trial protocol (RT-NOW). BMC Palliat Care. 2025 Apr 7;24(1):96. doi: 10.1186/s12904-025-01724-3. PMID 40189509